CLINICAL TRIAL: NCT01239095
Title: Perioperative Administration of Oral Green Tea Extract/Milk Thistle Extract to Colorectal Cancer Patients Undergoing Colorectal Cancer Resection, a Phase 1 Study
Brief Title: Oral Green Tea Extract and Milk Thistle Extract to Colorectal Cancer Patients Undergoing Resection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Richard Whelan (Other)
Collaborators: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor-Investigator, Richard Whelan, Professor, Feinstein Institute for Medical Research
Organization: Northwell Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-0002; 10-089 (Other: St Luke's Roosevelt)
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Green Tea and Milk Thistle Supplements (Experimental): Patients will receive green tea extract and milk thistle extract supplements for one week prior to surgery and for 30 days after surgery.
  Interventions: Drug: Green Tea and Milk Thistle Supplements

INTERVENTIONS:
Drug: Green Tea and Milk Thistle Supplements — Green Tea Extract: 3,200 mg per day Milk thistle extract with phosphatidylcholine: 2,700 mg per day
  Other Names: Green Tea Extract: EGCg; Milk Thistle Extract: Siliphos

SUMMARY:
Colorectal cancer is the third most common form of cancer found in the United States. To date surgical resection provides the best chance for cure. Unfortunately, despite "curative" surgery, tumor recurrences develop in 30-40% of patients from either unforeseen residual metastases or from viable tumor cells shed into the circulation before or at the time of surgery. There is evidence from both humans and mice suggesting that tumor growth is stimulated after surgery for a period of time.

This study calls for the administration of a green tea extract and a milk thistle extract, two orally ingested supplements, during the week immediately before and weeks after your surgery. It is not the current standard of care to give anti-cancer drugs during the perioperative period. The basic idea behind this study is that it should be beneficial to inhibit cancer growth in the days leading up to and following surgery. Why is this the case?

It makes sense to limit or inhibit tumor growth before surgery with drugs provided it can be done safely and does not interfere with the surgery. It is also logical to give anti-cancer drugs after surgery because, unfortunately, about 35 percent of colorectal cancer patients, after resection, have hidden tumor cells that remain in the body. There is also strong human evidence that tumor growth is stimulated during the first month after tumor resection as a result of the surgical injuries and the healing process. Therefore, there is good reason to give anti-cancer drugs as soon as possible after surgery in order to offset some of surgery's negative effects.

Although both supplements have been given safely to a wide variety of patients with a number of different medical problems, the two supplements together have never been given to cancer patients during the weeks just before and following surgery. The researchers hypothesize that the administration of these two supplements together will be safe in the period surrounding colorectal cancer surgery.

DETAILED DESCRIPTION:
Green tea extract and Silibinin (from the milk thistle plant) have both been shown in experimental studies to have anti-cancer effects as well as limited toxicity. Epigallocatechin-3-gallate (EGCG) is the major active catechin in green tea; it has been shown to prevent and limit tumor growth in murine models1-3. Silymarin, which is extracted from the seeds of the milk thistle plant, is used clinically as a hepatoprotective agent in Europe4. Its major active component, Silibinin, is well-tolerated and largely free of adverse effects5-6. In recent studies, Silibinin has been shown to inhibit the growth of a number of cancers in mouse models, including lung7, bladder8, liver9, prostate10, and colon11-12. Silibinin and EGCG have similar anti-neoplastic mechanisms including: 1) cell cycle arrest via upregulation of P21 and P27 and downregulation of CDK, 2) induction of apoptosis via Caspase-3 activation and cleavage of poly (ADP-ribose) polymerase (PARP), and 3) suppression of angiogenesis and metastasis via inhibition of vascular endothelial growth factor (VEGF) and matrix metalloproteinase (MMP-9)

ELIGIBILITY:
Inclusion Criteria:

* Patients must be age 18 to 85 years
* Patient must have biopsy proven colon or rectal cancer
* Cancer should be judged to be stage 1 to 3 based on preoperative staging
* Patients may be any race and any gender

Exclusion Criteria:

* Patients with cancer judged to be stage 4 are not eligible
* Patients undergoing emergency surgery for cancer are not eligible
* Patients who are immunosuppressed or taking immunosuppressive medications (steroids or chemotherapeutic agents) are not eligible
* Patients with Crohn's disease or ulcerative colitis are not eligible
* Patients with other malignancies are not eligible
* Patients who are taking part in other neoadjuvant and early adjuvant chemotherapy trials are not eligible

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-07; Primary Completion 2023-02 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events or complications | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Whelan, MD, Principal Investigator — Mount Sinai St. Luke's Roosevelt Hospital
Locations (1):
- Mount Sinai St. Luke's Roosevelt Hospital Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No